CLINICAL TRIAL: NCT04893213
Title: Socioeconomic Position and the Impact of Increasing the Proportion of Lower Energy Foods Available on Supermarket Meal Choices and Consumption
Brief Title: Increasing Availability of Lower Energy Meals on Food Choice and Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liverpool (Other)
Responsible Party: Principal Investigator, Eric Robinson, Reader in Psychological Sciences, University of Liverpool
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 8710 Ready Meal Menu Study
Record Dates: First submitted 2021-05-10; First posted 2021-05-19 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Diet, Healthy; Food Selection; Obesity; Eating Behavior
Keywords: availability; socio-economic position; food choice; eating behaviour
MeSH Terms: conditions — Food Preferences; Obesity; Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baseline availability (Active Comparator): Baseline availability of lower energy meal options
  Interventions: Other: Manipulation of availability of lower energy meal options
- Increased availability (Experimental): Increased availability of lower energy meal options
  Interventions: Other: Manipulation of availability of lower energy meal options

INTERVENTIONS:
Other: Manipulation of availability of lower energy meal options — Menus provided differ in % of menu options that are higher vs. lower in energy

SUMMARY:
This study will examine the effectiveness of a structural intervention (baseline proportion of lower energy ready meals vs increased proportion of lower energy ready meals) on calories (kcal) ordered and consumed. The study will use a within-subjects design, meaning all participants will be exposed to both conditions (baseline vs increased lower energy meal menus). The procedure will involve participants placing orders for supermarket ready meals, which are then delivered to their homes for their consumption. This study will also investigate whether the effectiveness of the intervention varies, depending on socioeconomic position (SEP). The primary hypothesis is that increasing proportion of lower energy options will decrease total kcal ordered and consumed, and that there will be no difference between higher and lower SEP. To address the limited evidence on longer term impacts of dietary interventions on daily energy intake, the present study will also examine post-meal energy consumption up to midnight on the following day. Finally, this study will explore the psychological processes that might underlie the effectiveness of the intervention among individuals with higher and lower SEP; namely, food choice motives, satiety responsiveness, plate clearing tendencies, and food waste concerns.

DETAILED DESCRIPTION:
See attached protocol documents.

ELIGIBILITY:
Inclusion Criteria:

* UK (United Kingdom) residents, aged 18 or over
* Fluent in English
* Have access to a phone/tablet/computer device which has access to Internet and a functioning camera
* Willing to consume two supermarket ready meals
* Have access to a functioning microwave and oven for the preparation of the ready meals

Exclusion Criteria:

* Taking part more than once
* Another member of the same household has participated in the study (Multiple members of the same household will not be allowed to take part)
* Current or historic diagnosed eating disorders
* Currently on any medication which affects appetite
* Any of the following dietary restrictions, intolerances, or allergies (Vegetarian, vegan, gluten-free, sugar-free, dairy/lactose-free, food allergy - such as milk, eggs, nut, wheat, fish, etc)
* History of severe childhood allergies, anaphylaxis or anaphylactic shock

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-04-13 (Actual); Primary Completion 2021-07-05 (Actual); Study Completion 2021-07-05 (Actual)

PRIMARY OUTCOMES:
Total meal energy (kcal) ordered | 20 minutes (the time frame denotes time taken to complete the initial study questionnaire and make the food choices)
  Calculated as the sum of the kcal content of the main and side ordered
Total meal energy (kcal) consumed | Once the food has been delivered, the time frame is up to 72 hours
  Calculated as the sum of the kcals consumed from the main and side combined

SECONDARY OUTCOMES:
Post-meal intake (kcal) | Measured 24-30 hours after study meal is consumed
  Calculated as total energy (kcal) consumed after the study meal until midnight on the following day (dietary recall).

CONTACTS AND LOCATIONS:
Overall Officials: Eric Robinson, PhD, Principal Investigator — Study Principal Investigator
Locations (1):
- University of Liverpool, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Shared on the Open Science Framework (OSF)
Supporting Information: Study Protocol, SAP
Time Frame: On publication, indefinitely
Access Criteria: Open website
URL: https://osf.io/yku5q/

REFERENCES:
- Available data/document: Study Protocol — https://osf.io/yku5q/ — Protocol on the Open Science Framework (OSF)
- Available data/document: Statistical Analysis Plan — https://osf.io/yku5q/
- Available data/document: Individual Participant Data Set — https://osf.io/yku5q/ — The study protocol and statistical analysis plan were pre-registered on the OSF prior to starting recruitment. IPD will be made available when results are published.